CLINICAL TRIAL: NCT05505175
Title: TREATMENT PATTERNS AND CLINICAL OUTCOMES AMONG PATIENTS IN BRAZIL RECEIVING PALBOCICLIB COMBINATIONS FOR HR+/HER2- ADVANCED/METASTATIC BREAST CANCER IN REAL WORLD SETTINGS
Brief Title: Outcomes Among Patients in Brazil Receiving Palbociclib Combinations for HR+/HER2- MBC
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481168; IRIS Brazil (Other: Alias Study Number)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Breast Carcinoma
Keywords: non-metastatic breast cancer; locally advanced (stage III) breast cancer; metastatic breast cancer (stage IV)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Breast Cancer Patients: Eligible patients including patients with a potential follow-up period of 6 months following the index date

SUMMARY:
The objective of this study is to describe patient demographics, clinical characteristics, treatment patterns and clinical outcomes of adult female patients who have received palbociclib combination treatments as first line therapy, regardless of combination partner and labelled use in real world settings across Brazil.

DETAILED DESCRIPTION:
The primary objective of this real world study is to describe patient demographics, clinical characteristics, treatment patterns and clinical outcomes of adult female patients who have received palbociclib combination treatments as first line therapy, regardless of combination partner and labelled use.

Primary Objectives

* To describe the demographic and clinical characteristics of patients who have received palbociclib combination treatments in line with locally approved indications.
* To describe adjuvant therapies received for their treatment of early or locally advanced breast cancer (Stages 0-IIIa).
* To describe treatments received in the advanced/metastatic setting, before and after palbociclib combination use.
* To describe dosing and dose changes, interruptions, delays, and discontinuations associated with palbociclib use in clinical practice.
* To describe supportive therapies received by patients while receiving palbociclib combination treatments.
* To determine the following outcome in overall population and defined subgroups for patients who had received palbociclib combination treatment for at least 6 months:

  * Progression-free survival;
  * Objective response rate (ORR);
  * Proportion of patients alive.

Exploratory Objectives

• To evaluate progression-free survival (PFS) associated with palbociclib combination treatments after 1 and 2 years following Palbociclib combination treatment.

This study will be conducted as a retrospective medical record review of patients who have received palbociclib combination treatments as first line treatment regardless of combination. The study will comprise of a medical record review conducted in Brazil. The study design is similar to a previously conducted RWE IRIS Global study previously conducted in multiple other countries (protocol no. A5481090) .

Data collection will be online via electronic data capture using electronic case report form (eCRF). Each physician will be asked to select all the medical records of approximately 5-20 patients per site (approximate total: 300 patients) who meet the inclusion criteria and then invited to complete the eCRF from each enrolled patient. Time to complete each eCRF will be 30 minutes, approximately.

In order to allow for a sufficiently long observational window, physicians will be asked to go back to a specific point in time, the index date, and sequentially select the medical records of the next 'n' patients who meet the inclusion criteria. The 'index date' will be defined as 30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil (eg, if palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole the next day, the index date will be April 2, 2018).

The advantage to a retrospective medical record review approach over a database analysis is that of being designed specifically to collect data that fulfils the study objectives. Thus, it readily collects and informs on all key drug related clinical outcome measures of critical importance to this study, in a consistent manner, across countries if reported in a medical record. The resulting data set enables direct comparisons across markets, delivering in turn greater confidence in the reliability of conclusions drawn from the research. An additional advantage of this approach lies in the ability to obtain information that only the treating physician may be aware of, such as the reasons for treatment switches or discontinuations or more perceptive questions that rely on the physician's professional opinion.

ELIGIBILITY:
Inclusion Criteria:

* HR+/HER2- breast cancer diagnosis with confirmed ABC/MBC
* Received palbociclib as a first line therapy
* No prior or current enrolment in an interventional clinical trial for ABC/MBC
* Have a potential follow-up period of 6 months following the index date (30 days after first palbociclib prescription: palbociclib with fulvestrant and/or palbociclib with letrozole/aromatase inhibitor).

Exclusion Criteria:

* Patients who were enrolled to receive fulvestrant but already received previous therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants only
Study Population: Adult female patients with HR+/HER2 non-metastatic breast cancer who progressed to locally advanced (stage IIIB/C) or metastatic (stage IV) breast cancer receiving palbociclib combination regimens as per the approved indication.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Demographical characteristics of patients who have received palbociclib combination treatments in line with locally approved indications | 30 days after prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Adjuvant treatments received for subset of patients previously diagnosed with non-metastatic breast cancer who progressed to locally advanced (stage IIIB/C) or metastatic (stage IV) breast cancer. | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe treatments received in the advanced/metastatic setting before palbociclib combination use | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe treatments received in the advanced/metastatic setting after palbociclib combination use | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe dosing associated with palbociclib use in clinical practice | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe dose changes associated with palbociclib use in clinical practice | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe interruptions associated with palbociclib use in clinical practice | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe delays associated with palbociclib use in clinical practice | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe discontinuations associated with palbociclib use in clinical practice | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Describe supportive therapies received by patients while receiving palbociclib combination treatments | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Proportion of patients who are progression free following clinical outcomes in overall population and defined subgroups for patients who had a potential follow-up of 6 months after palbociclib combination treatment initiation | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Real world Objective response rate (ORR) following clinical outcomes in overall population and defined subgroups for patients who had a potential follow-up of 6 months after palbociclib combination treatment initiation | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.
Proportion of patients alive following clinical outcomes in overall population and defined subgroups for patients who had a potential follow-up of 6 months after palbociclib combination treatment initiation | 30 days after the physician first prescribed palbociclib + partner therapy until completion of this study in 2022.
  30 days after the physician first prescribed palbociclib + partner therapy following the approval of the indication in Brazil . From when palbociclib + letrozole was available Feb 1, 2018 in Brazil and the physician initiated a patient on palbociclib+ letrozole until completion of this study in 2022.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Brazil (14):
  - NOB - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Ensino E Terapia de Inovação Clínica Amo - Ética, Salvador, Estado de Bahia
  - Instituto D´Or de Pesquisa E Ensino - Brasília, Brasília, Federal District
  - Hospital Sírio Libanês, Brasília, Federal District
  - Hospital Araújo Jorge, Goiânia, Goiás
  - Oncoclínicas Do Brasil Servicos Médicos S/A - Oncocentro, Belo Horizonte, Minas Gerais
  - Centro Especializado de Oncologia de Florianópolis, Florianópolis
  - Instituto de Mastologia e Oncologia, Goiânia
  - Instituto D'or de Pesquisa e Ensino, Recife
  - Centro de Tratamento de Tumores Botafogo, Rio de Janeiro
  - Instituto D´or de Pesquisa e Ensino, Rio de Janeiro
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - Hospital Paulistano - INSTITUTO DE EDUCAÇÃO, PESQUISA E GESTÃO EM SAÚDE, São Paulo
  - Hcor - Associação Beneficente Síria, São Paulo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481168